CLINICAL TRIAL: NCT03183037
Title: Acupuncture for Persistent Chemotherapy-induced Peripheral Neuropathy Symptoms in Solid Tumor Survivors: A Pilot Study
Brief Title: Acupuncture for Symptoms of Nerve Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-298
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Peripheral Neuropathy; Chemotherapy-induced Peripheral Neuropathy
Keywords: Acupuncture; 17-298
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Acupuncture Therapy; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Three - arm pilot randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture Treatment Group (Experimental): Ten acupuncture treatments over the course of eight weeks, with twice weekly acupuncture treatments for the first two weeks, and then weekly treatment thereafter.
  Interventions: Procedure: Acupuncture; Behavioral: questionnaires
- Sham Acupuncture Treatment Group (Placebo Comparator): Ten sham acupuncture treatments over the course of eight weeks, with twice weekly sham acupuncture treatments for the first two weeks, and then weekly sham acupuncture treatment thereafter.
  Interventions: Procedure: Sham Acupuncture; Behavioral: questionnaires
- Usual Care Group (Active Comparator): Twelve weeks of usual care.
  Interventions: Other: Usual Care Group; Behavioral: questionnaires

INTERVENTIONS:
Procedure: Acupuncture — The acupuncture group will undergo 8 weeks of outpatient acupuncture or sham acupuncture treatments (twice weekly for 2 weeks, then weekly for 6 weeks, 10 treatments in total). The investigators have designed this approach to standardize acupuncture treatment for future broad use; it is based on the understanding that CIPN is a global symptom complex rather than individual isolated or local symptoms.
  Arms: Acupuncture Treatment Group
Procedure: Sham Acupuncture — Subjects in this group will receive the sham acupuncture procedure on the same schedule as subjects in the real acupuncture group. In both groups, patients' eyes will be covered with patches so they cannot observe the treatment procedure. To improve incentive to join and stay in the study, we will unblind all patients at Week 12, and offer those randomized to the Sham group 8 weeks of Acu (real) treatment. All points used will be documented.
  Arms: Sham Acupuncture Treatment Group
Other: Usual Care Group — Patients go to clinic three times during the study, at Baseline, Week 8, and Week 12 to undergo QST and CPM tests. Patients will complete all questionnaires (CIPN severity by 0-10 11-point numeric rating scale, FACT/GOG-Ntx-11, NPS) and their pain medication use at these time points. Week 4 questionnaires can be completed over the phone. As an incentive for patients to join the study - and for those randomized to control to stay in the study - controls will be offered 8 weeks of Acu (real) treatment once they have completed Week 12 assessments.
  Arms: Usual Care Group
Behavioral: questionnaires — FACT/GOG-Ntx, Neuropathic Pain Scale (NPS),Treatment Expectancy Scale (TES), Quantitative Sensory Testing (QST), Insomnia Severity Index (ISI), Hospital Anxiety and Depression Scale (HADS), Brief Fatigue Inventory (BFI)

SUMMARY:
The purpose of this study is to compare the effects of real acupuncture with placebo acupuncture or usual care on symptoms of nerve damage from chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age ≥ 18 years old
* Solid tumor survivors with no evidence of disease
* Moderate to severe CIPN, defined by symptoms such as numbness, tingling, or pain ratings of 4 or greater on a 0-10 numeric rating scale (NRS)
* Have completed neurotoxic chemotherapy at least 3 months prior to enrollment
* If taking anti-neuropathy medications, they are on a stable regimen (no change in 3 months)

Exclusion Criteria:

* Patients with a pacemaker
* Prior acupuncture treatment within 5 years of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
change in the proportion of patients with a CIPN severity | up to 12 weeks
  according to the NCI-CTC 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Ting Bao, MD, DABMA, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhi WI, Baser RE, Talukder D, Mei YZ, Harte SE, Bao T. Mechanistic and thermal characterization of acupuncture for chemotherapy-induced peripheral neuropathy as measured by quantitative sensory testing. Breast Cancer Res Treat. 2023 Feb;197(3):535-545. doi: 10.1007/s10549-022-06846-3. Epub 2022 Dec 17. PMID 36527520
- [Derived] Zhi WI, Chen P, Kwon A, Chen C, Harte SE, Piulson L, Li S, Patil S, Mao JJ, Bao T. Chemotherapy-induced peripheral neuropathy (CIPN) in breast cancer survivors: a comparison of patient-reported outcomes and quantitative sensory testing. Breast Cancer Res Treat. 2019 Dec;178(3):587-595. doi: 10.1007/s10549-019-05416-4. Epub 2019 Aug 27. PMID 31456070
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm